CLINICAL TRIAL: NCT05170269
Title: Prevention of Maternal-fetal Cytomegalovirus Transmission After Primary Maternal Infection With Gestational Age ≤ 14 Weeks - an Open-label, Single-arm, Prospective Trial Investigating Efficacy and Safety of Cytotect CP Biotest
Brief Title: Prevention of Maternal-fetal Cytomegalovirus Transmission After Primary Maternal Infection, GW ≤ 14 (PreCyssion)
Acronym: PreCyssion
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Biotest (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 997; 2020-002383-32 (EudraCT Number)
Record Dates: First submitted 2021-10-19; First posted 2021-12-27 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-12

CONDITIONS: Congenital Cytomegalovirus Infection
Keywords: Cytomegalovirus; Pregnancy; CMVIG; maternal CMV infection
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BT097 (Experimental): Subjects will receive BT097 200 U per kg of maternal body weight intravenously every 2 weeks until at least GW 17
  Interventions: Drug: BT097

INTERVENTIONS:
Drug: BT097 — Subjects will receive BT097 200 U per kg of maternal body weight intravenously every 2 weeks until at least GW 17
  Other Names: Cytotect CP Biotest 100 U/mL solution for infusion

SUMMARY:
A phase 3, open-label, single-arm, prospective, multi-center trial of Cytotect CP Biotest (BT097) for prevention of maternal-fetal CMV transmission after primary maternal CMV infection. The main purpose of the trial is to demonstrate efficacy and safety of Cytotect CP Biotest in preventing maternal-fetal transmission of cytomegalovirus (CMV).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from subjects indicating that they understand the purpose of and procedures required for the trial and are willing to participate in it
* Pregnant women, age 18 to 45 years
* Pregnant women at trial entry with gestational age ≤14 weeks; pregnancy after in-vitro fertilization permitted
* Detection of early primary CMV infection

Exclusion Criteria:

* Women with current multiple pregnancy
* History of severe pre-eclampsia or severe gestational hypertension (GHTN), which required medical intervention. Definition according to AWMF guideline (AWMF, 2019)
* Presence of severe disease impairing course of pregnancy (e.g. diabetes, epilepsy, cancer)
* Congenital or acquired autoimmune disease
* Known immunosuppressive (e.g., transplanted patients) or immunodeficient condition
* Known infection with hepatitis B or C, or HIV from the medical history or active infection at screening as assessed by respective virus serology
* Maternal CMV infection prior to this pregnancy (preconceptional CMV infection)
* Covid-19 infection at time of inclusion
* Any signs or symptoms indicating an increased risk of abortion or premature labor or has known negative effect on fetus with exception of a CMV infection
* Active infection according to TORCH serology with exception of CMV in the assessment of the investigator
* Known major fetal anomalies or demise
* Intolerance to proteins of human origin or known allergic reactions to components of the trial product
* Selective absolute IgA deficiency or known antibodies to IgA
* Known pre-existing clinically relevant risk factors for thrombotic events
* Known renal insufficiency with serum creatinine levels >1.4 mg/dL and proteinuria (albuminuria) at screening (≥30 mg/dL or dipstick reading of 1+ and greater)
* Participation in another clinical trial within 90 days before entering the trial or during the trial
* Women who are dependent on trial site staff, on Biotest AG or its authorized representatives
* Inability or lacking motivation to participate in the trial
* Medical condition, laboratory finding, or physical examination finding that in the opinion of the investigator precludes participationInability or lacking motivation to participate in the trial
* Eligibility for a subgroup where enrollment was stopped

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 48 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2023-11-19 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
To determine the overall rate of maternal-fetal transmission at the time of amniocentesis (week 20 [-1 week / +2 weeks] of gestation) | Gestational week 19 - week 22
  To determine the overall rate of maternal-fetal transmission at the time of amniocentesis

SECONDARY OUTCOMES:
Subgroups: (1) Subjects with periconceptionally acquired infection or (2) Subjects with infection acquired during first trimester | Gestational week 20 +-1 Week
  To determine the rate of maternal-fetal transmission at the time of amniocentesis
To determine maternal CMV viral load (copies/ml) | until gestational week 30
  Number of CMV-DNA copies (copies/mL) and corresponding absolute and percentage changes from baseline, until gestational week (GW) 30
To determine maternal anti-CMV IgG Levels (U/ml) | until gestational week 30
  Maternal anti-CMV IgG Levels (U/ml), absolute and percentage changes from baseline
To determine maternal anti-CMV IgG avidity (%) | until gestational week 30
  Number/percentage of subjects with Low, Intermediate, High avidity
To determine maternal anti-CMV IgM index (Index) | until gestational week 30
  Number/percentage of subjects with non-reactive, indeterminate and reactive cut-off index (COI)
To determine soluble fms-like tyrosine kinase 1 (sFlt-1) concentration in maternal serum | until gestational week 30
  Number/percentage of subjects with high (≥1504 pg/mL) or low (<1504 pg/mL) values
To evaluate vitality of the fetuses/newborns | until date of delivery
  Number/percentage of subjects with Normal / Abnormal Not Clinically Significant / Abnormal Clinically Significant results per parameter and visit
To evaluate growth of the fetuses/newborns | Until date of delivery
  Number/percentage of subjects with Normal / Abnormal Not Clinically Significant / Abnormal Clinically Significant results per parameter and visit
To evaluate the rate of congenital CMV infection at delivery or within the first 3 days after delivery | Date of Delivery + 3 days
  To evaluate the rate of congenital CMV infection at delivery or within the first 3 days after delivery
To measure the number of CMV-DNA copies in the urine of newborns | Date of Delivery
  To measure the number of CMV-DNA copies in the urine of newborns
To assess the number, severity, causality, outcome, and seriousness of all adverse events (AEs)/ treatment-emergent AEs (TEAEs)/ AEs of special interest until delivery (+3 days) in both mother and fetus/newborn | Date of Delivery + 3 days
  To assess the number, severity, causality, outcome, and seriousness of all adverse events (AEs)/ treatment-emergent AEs (TEAEs)/ AEs of special interest until delivery (+3 days) in both mother and fetus/newborn

CONTACTS AND LOCATIONS:
Overall Officials: Karl O Kagan, Prof, Principal Investigator — Universitätsklinik Tuebingen - Frauenklinik; 72076 Tübingen
Locations (5):
- Germany (5):
  - 4906, Berlin
  - 4903, Bonn
  - 4902, Erlangen
  - 4901, Tübingen
  - 4905, Wasserburg am Inn